CLINICAL TRIAL: NCT04349800
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of KVD900 Followed by Crossover Sub-studies of KVD900 Formulations, and Food Effect in Healthy Male Volunteers
Brief Title: A Single Dose Safety, Tolerability, Pharmacokinetic and Food Effect Study of KVD900 (Sebetralstat) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KVD900-101
Record Dates: First submitted 2020-03-09; First posted 2020-04-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Angioedema
Keywords: Sebetralstat
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Single Ascending Dose - 5 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Single Ascending Dose - 10 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Single Ascending Dose - 20 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Single Ascending Dose - 40 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Single Ascending Dose - 80 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Single Ascending Dose - 160 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Single Ascending Dose - 300 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Single Ascending Dose - 600 mg (Experimental)
  Interventions: Drug: KVD900; Drug: Placebo to KVD900
- Formulation Screen (Experimental)
  Interventions: Drug: KVD900
- Food Effect (Experimental)
  Interventions: Drug: KVD900

INTERVENTIONS:
Drug: KVD900 — Active
Drug: Placebo to KVD900 — Placebo
  Arms: Single Ascending Dose - 10 mg; Single Ascending Dose - 160 mg; Single Ascending Dose - 20 mg; Single Ascending Dose - 300 mg; Single Ascending Dose - 40 mg; Single Ascending Dose - 5 mg; Single Ascending Dose - 600 mg; Single Ascending Dose - 80 mg

SUMMARY:
A safety, tolerability, pharmacokinetic and food effect study of KVD900 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 55 years of age.
* Healthy subjects as determined by past medical history and as judged by the Chief Investigator or designee.
* Male subject willing to use a highly effective method of contraception.
* Subject with a body mass index (BMI) of 18-32 kg/m2.
* Subject with no clinically significant history of previous allergy or sensitivity to KVD900 or any of the excipients contained within the investigational medicinal product (IMP).
* Subject with no clinically significant abnormal serum biochemistry, haematology, clotting profiles, and urine examination values within 28 days before the first dose of IMP.
* Subject with a negative urinary drugs of abuse screen, determined within 28 days before the first dose of IMP
* Subject with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
* Subject with no clinically significant abnormalities in 12-lead electrocardiogram
* Subjects must not donate sperm from first dose until at least 3 months after last dose of IMP.
* Subjects without any special food restrictions that would hinder ability to consume the high fat breakfast provided during study Part C; such as lactose intolerance , vegan, low-fat, low sodium, etc.
* Subjects with no known allergy or sensitivity to lactose and/or any additional excipients contained in IMP.
* Subject must be available to complete the study (including all follow up visits).
* Subject must satisfy the Chief Investigator or designee about their fitness to participate in the study.
* Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence IMP absorption.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements .
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular (no history of syncope or vasovagal events), or metabolic dysfunction.
* Subjects with a history of clotting abnormalities.
* A clinically significant history of drug or alcohol abuse in the last 5 years.
* Users of nicotine products i.e., current smokers or ex-smokers who have smoked within the 6 months prior to dosing with the study medication or users of cigarette replacements.
* Inability to communicate well with Investigators.
* Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of IMP.
* Donation of 450 mL or more blood within the 3 months before the first dose of IMP.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events | Change from pre-dose to last visit, 5-7 days post dose.
Number of Subjects with Serious Adverse Events | Change from pre-dose to last visit, 5-7 days post dose.
Number of participants with clinically significant changes in laboratory assessments | Throughout study until last visit, 5-7 days post dose.
Number of participants with clinically significant changes in vital signs | Throughout study until last visit, 5-7 days post dose.
Number of participants with clinically significant changes in electrocardiogram (ECG) measurements | Throughout study until last visit, 5-7 days post dose.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | Up to 48 hours post dose
  Derived from time-concentration plasma levels of KVD900
Pharmacokinetics - AUC0-t | Up to 48 hours post dose
  Derived from time-concentration plasma levels of KVD900
Pharmacokinetics - AUC0-24 | Up to 24 hours post dose
  Derived from time-concentration plasma levels of KVD900
Pharmacokinetics - AUC0-inf | Up to 48 hours post dose
  Derived from time-concentration plasma levels of KVD900
Pharmacokinetics - food effect (Part C only) | Up to 24 hours post dose
  90% confidence intervals of the ratios for AUC0-t and Cmax with and without food lie in the range 80-125
Pharmacokinetics - formulation bridge - relative bioavailability (Part B only) | Up to 24 hours post dose
  90% confidence intervals of the ratios for AUC0-t and Cmax between the two dosages lie in the range 80-125

CONTACTS AND LOCATIONS:
Locations (1):
- KalVista Investigative Site, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maetzel A, Smith MD, Duckworth EJ, Hampton SL, De Donatis GM, Murugesan N, Rushbrooke LJ, Li L, Francombe D, Feener EP, Yea CM. KVD900, an oral on-demand treatment for hereditary angioedema: Phase 1 study results. J Allergy Clin Immunol. 2022 Jun;149(6):2034-2042. doi: 10.1016/j.jaci.2021.10.038. Epub 2022 Jan 24. PMID 35086692